CLINICAL TRIAL: NCT03970850
Title: Multi-Center Clinical Performance Evaluation of the NeuMoDx™ Chlamydia Trachomatis (CT) / Neisseria Gonorrhoeae (NG) [CT/NG] Assay on the NeuMoDx™ 288 Molecular System and the NeuMoDx™96 Molecular System
Brief Title: NeuMoDx PrEDiCTiNG Study Evaluation Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuMoDx Molecular, Inc. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTNG-01-18NMD
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Chlamydia Trachomatis Infection; Neisseria Gonorrheae Infection
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Multi-arm - Symptomatic and Asymptomatic Males (Active Comparator): Arm 1 - Urine from males subjects
  Interventions: Diagnostic Test: NeuMoDx CT/NG Assay
- Multi-arm - Symptomatic and Asymptomatic Females (Active Comparator): Arm 2 - Endocervical, self-collected (in the clinical setting) and physician-collected vaginal swabs and urine from female subjects
  Interventions: Diagnostic Test: NeuMoDx CT/NG Assay
- Multi-arm - FDA cleared NAATs (Comparator) (Active Comparator): Arm 3 - Comparator (for females - vaginal and urine NAATs and for males - 3 urine NAATs)
  Interventions: Diagnostic Test: FDA-cleared NAATs

INTERVENTIONS:
Diagnostic Test: NeuMoDx CT/NG Assay — NeuMoDx CT/NG Assay as implemented on NeuMoDx 288 Molecular System and NeuMoDx 96 Molecular System
  Arms: Multi-arm - Symptomatic and Asymptomatic Females; Multi-arm - Symptomatic and Asymptomatic Males
Diagnostic Test: FDA-cleared NAATs — Testing swabs and urine specimen from both male and female subjects on the FDA-cleared NAATs
  Arms: Multi-arm - FDA cleared NAATs (Comparator)

SUMMARY:
This investigational study will be conducted to evaluate the performance of the NeuMoDx™ CT/NG Assay on the NeuMoDx™ 288 Molecular System and NeuMoDx™ 96 Molecular System (collectively referred to as NeuMoDx™ CT/NG Assay test system).

DETAILED DESCRIPTION:
Clinical performance characteristics of the NeuMoDx CT/NG Assay on NeuMoDx™ 288 Molecular System and NeuMoDx™ 96 Molecular System will be evaluated in a multi-center, prospective, sampling study by comparing the diagnoses made by the NeuMoDx™ CT/NG Assay to Patient Infected Status (PIS) as the reference standard.

Prospectively collected urine and swab specimens from individual subjects will be tested using the NeuMoDx™ CT/NG Assay at one of the three NeuMoDx testing sites. Subjects' PIS for CT and PIS for NG will be determined by a central laboratory using FDA-cleared, legally marketed CT/NG combo assays on pre-specified sample matrices according to the PIS determination algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects of at least 14 years of age or older.
2. Subject must be able and willing to provide informed consent. The use of a 'surrogate' or 'Legally Authorized Representative' is allowed and shall follow the site's standard procedures, under which the clinical investigation will be conducted.
3. Subjects undergoing a routine pelvic examination, subjects eligible for screening evaluations for possible STDs and/or subjects known to be partners with a person with a confirmed or suspected STD.
4. Subject is willing to provide all required specimens.

Exclusion Criteria:

1. Female subject reports that she had a hysterectomy.
2. Subject self-reports use of antibiotics within 28 days of study enrollment.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Subjects eligible for CT/NG screening (make sure it matches the protocol)
Enrollment: 4017 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Clinical specificity and sensitivity | Through study completion, an average of 1 year
  Clinical specificity and sensitivity of NeuMoDx CT/NG Assay for both CT and NG relative to an individual's patient infected status (PIS)

SECONDARY OUTCOMES:
Valid results rate | Through study completion, an average of 1 year
  Evaluate indeterminate and unresolved rates

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - Healthcare Clinical Date, Inc. (Segal Trials), North Miami, Florida
  - Planned Parenthood - Southwest and Central Florida, Orlando, Florida
  - Planned Parenthood - Southwest and Central Florida, Tampa, Florida
  - Indiana University (IU), Indianapolis, Indiana
  - LSU Health Science, New Orleans, Louisiana
  - NeuMoDx Molecular, Inc., Ann Arbor, Michigan
  - Henry Ford Health System (HFHS), Detroit, Michigan
  - Planned Parenthood - Northern, Central and Southern New Jersey, Elizabeth, New Jersey
  - Planned Parenthood - Northern, Central and Southern New Jersey, Newton, New Jersey
  - Planned Parenthood - Northern, Central and Southern New Jersey, Riverside Park, New Jersey
  - TriCore Reference Labs, Albuquerque, New Mexico
  - MetroHealth Medical Center, Cleveland, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Planned Parenthood - Gulf Coast, Houston, Texas

IPD SHARING:
Plan to Share IPD: No